CLINICAL TRIAL: NCT04224389
Title: Prospective Non-randomized Comparative Study Between IMRT and Primary Transoral Surgery in the Treatment of Squamous Cell Carcinomas of Early Local Stage of Oropharynx
Brief Title: IMRT and Primary Transoral Surgery in the Treatment of Squamous Cell Carcinomas
Acronym: TORPHYNX
Status: Recruiting | Type: Observational
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-A02253-50; 2017/2617 (Other: CSET number (Gustave Roussy ID))
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Squamous Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Radiotherapy: IMRT on the primitive site and the lymph nodes. +/- Concomitant chemotherapy at the discretion of the meeting multidisciplinary
  Interventions: Radiation: IMRT
- Surgery: transoral resection of the primary tumor, with cervical lymph node dissection. Radiotherapy complementary according to the histological criteria of severity
  Interventions: Procedure: transoral resection

INTERVENTIONS:
Procedure: transoral resection — The technique of transoral surgery will be left to the choice of the surgeon according to the equipment and the experience of the team and will be gathered. The options are: transoral surgery robot-assisted, endoscopic laser transoral surgery, transoral laser surgery classical instruments. The exact description of the resected area will be collected. of the cross-sections will be made for extemporaneous analysis if necessary in lateral margins and deep until complete excision.
  Groups: Surgery
Radiation: IMRT — Intensity modulation radiotherapy (RCMI or IMRT) will be performed using techniques static or rotational (arctherapy, tomotherapy). Restraint is recommended with thermoformed mask
  Groups: Radiotherapy

SUMMARY:
Compare patients' feelings in terms of swallowing ability assessed by the overall score of MD Anderson Dysphagia Inventory (MDADI) 2 years after starting treatment between patients who have been treated with IMRT and those who were treated by transoral surgery for a squamous cell carcinoma of the early stage oropharynx.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. ECOG performance status 0-2
3. Histologically confirmed squamous cell carcinoma
4. Primitive localization of the oropharynx on the tonsil compartment or the tongue base
5. p16 or HPV status available
6. TNM classification AJCC7th T1 or T2
7. TNM classification AJCC7th N0 or N1
8. Patient and tumor that can be treated by radiotherapy or by transoral surgery
9. Patient who has not objected to participate after being informed about the study. The patient must be able and willing to cooperate in follow-up and study visits

Exclusion Criteria:

1. Severe medical comorbidity or other contraindication to radiotherapy or surgery
2. Primary tumor or unresectable lymphadenopathy
3. Metastatic disease
4. History of squamous cell carcinoma of the head and neck within 5 years
5. History of radiation therapy to the head and neck
6. Inability to undergo or complete radiation therapy follow-up consultations
7. History of cancer except free of any disease for at least 5 years, with the exception of non-melanoma skin cancers
8. Inability to complete questionnaires
9. Pregnant or lactating woman
10. Patient under tutorship or curatorship, deprived of liberty or unable to do so to express consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who have been treated with IMRT and those who were treated by transoral surgery for a carcinoma squamous cell of the early stage oropharynx
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-06-22 (Actual); Primary Completion 2031-06 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
MD Anderson Dysphagia Inventory (MDADI) global score | 2 years after inclusion
  Score goes from 20 to 100. A higher score means a better ability to swallow

CONTACTS AND LOCATIONS:
Locations (16):
- France (16):
  - Gustave Roussy, Villejuif, Val De Marne
  - Centre Hospitalier InterCommunal, Créteil
  - Centre Oscar Lambret, Lille
  - Hôpital la Croix Rousse, Lyon
  - Centre Léon Bérard, Lyon
  - CHU Conception, Marseille
  - CHU Montpellier, Montpellier
  - CHU Nantes - Hôtel Dieu, Nantes
  - Institut Universitaire de la face et du cou, Nice
  - Hôpital Européen Georges Pompidou, Paris
  - CHU Reims, Reims
  - Hôpital Charles Nicolle, Rouen
  - CHU Hôpital de Hautepierre, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - CHU Tours, Tours
  - CHRU Nancy - Hôpital de Brabois, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: Yes